CLINICAL TRIAL: NCT00137228
Title: The Reliability and Concurrent Validity of the Figure-of-Eight Method of Measuring Hand Edema in Patients With Burn Injuries
Brief Title: Measuring Hand Edema in Burn Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Institute of Surgical Research (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-04-030
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2008-01-08 (Estimated); Status verified 2007-12

CONDITIONS: Edema
Keywords: Hand Edema; Figure of eight method; Measuring edema in burn patients
MeSH Terms: conditions — Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: figure-of-eight hand measurements
Procedure: water volumetry hand measurements

SUMMARY:
The purpose of this study is to determine the reliability and concurrent validity of the figure-of-eight method of measuring hand edema in the burn patient population. Establishing the reliability and validity would enable a more time efficient assessment than the currently accepted methods.

DETAILED DESCRIPTION:
A prospective study involving 33 burn patients admitted to the US Army Burn Center. Two raters will perform three separate blinded measurements for hand edema using the figure-of-eight measurement technique. A third rater will then perform two blinded measurements using water volumetry. All measurements will be read and recorded by an independent recorder. The three measurements of rater 1 and 2 will be analyzed to determine intratester reliability. The average of the three figure-of-eight measurements will be compared to measure intertester reliability. The two volumetry measurements will be compared to determine intratester reliability. The average of the 2 volumetry measurements and the average fo the three figure-of-eight measurements will be used to determine concurrent validity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-89 years old
* Admitted to the United States (U.S.) Army Burn Intensive Care Unit (ICU) or ward with burn injury and the presence of bilateral or unilateral hand edema

Exclusion Criteria:

* Subject unable to be placed in test position for volumetry testing or the presence of a medical condition, as defined by a physician, that precludes the safe use of volumetry.
* Subject is unable to tolerate his/her hand(s) being immersed in room temperature water for volumetry testing.
* Subject does not have any of the bony landmarks (due to amputation, previous surgery) required to perform the figure-of-eight measurement

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-01; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
The figure-of-eight method for measuring hand edema in burn patients is just as reliable and valid as water volumetry measurement. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Scott Dewey, PT, CHT, OCS, Principal Investigator — US Army Institute of Surgical Research
Locations (1):
- U.S. Army Institute of Surgical Research, Fort Sam Houston, Texas, United States

REFERENCES:
- [Background] Leard JS, Breglio L, Fraga L, Ellrod N, Nadler L, Yasso M, Fay E, Ryan K, Pellecchia GL. Reliability and concurrent validity of the figure-of-eight method of measuring hand size in patients with hand pathology. J Orthop Sports Phys Ther. 2004 Jun;34(6):335-40. doi: 10.2519/jospt.2004.34.6.335. PMID 15233395